CLINICAL TRIAL: NCT05303350
Title: Multicentric Study of Comparison of the Effectiveness of a Web Fracture Liaison Service (e_FLS) to Fracture Liaison Services in France: the evAB Study
Brief Title: Comparison of the Effectiveness of a Web Fracture Liaison Service (e_FLS) to Fracture Liaison Services in France: the evAB Study (evAB)
Acronym: evAB
Status: Withdrawn | Type: Observational
Why Stopped: logistic difficulties
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: French Society of Rheumatology (Other); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP211339; 2022-A00553-40 (Other: ID-RCB Number)
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Osteoporosis; Fracture
Keywords: Osteoporosis; Fracture; Fracture liaison service; Digital medicine
MeSH Terms: conditions — Osteoporosis; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- e_FLS: Patients detected by an automated patient detection tool with a web-based platform
- FLS: Control group / Conventional group : Patients followed in a conventional fracture liaison department

SUMMARY:
The purpose of this study is to compare web FLS model (e_FLS) to conventional FLS in terms of increasing the proportion of patients receiving an antiosteoporotic treatment in the year after a low trauma fracture.

DETAILED DESCRIPTION:
Osteoporotic fractures such as hip fractures and severe fractures are associated with increased morbidity and mortality and impose a large financial burden on healthcare systems. Patients with osteoporosis-related fractures are at higher risk of subsequent fractures. Other severe fractures (pelvis, vertebrae, humerus) have similar consequences, pelvis. The risk of refracture after fracture depends on the time: it is 5 times higher in the first 2-3 years, and 2 times higher after. This notion of Imminent Fracture Risk is the basis for the development of post-fracture care pathways called "fracture liaison. The implementation of FLS is the most effective way to reduce the risk of secondary fracture. Despite their success, FLS programs are not an integral part of post-fracture care throughout the France. The investigators believe that the barriers to the implementation of such a pathway are multiple and are largely related to the lack of accessibility for patients to FLS, and to the mobilization of important and unsustainable human resources. Some French public hospitals or institutions are currently building some e_FLS models based on an automatic detection of patients with fractures, and a on a cloud-based system where practitioners across the health care sector can communicate and jointly manage osteoporotic patients. The investigators' hypothesis is that this web FLS (e_FLS) is at least as effective as the classical FLS for the secondary fracture prevention.

The objective of the investigators' study is to compare web FLS model (e_FLS) to conventional FLS in terms of increasing the proportion of patients receiving an antiosteoporotic treatment in the year after a low trauma fracture (evAB project).

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged above 60 years, living in France, with fragility fractures in response to low-energy trauma (e.g., a fall from standing height).
* The patient or his legal representative does not object to the patient's participation in the research Note: Patients in guardianship or curatorship can be included in this protocol

Exclusion Criteria:

* Pathological fractures, high trauma fractures and per prosthetic fractures.
* Non registration with a social security scheme (holder or beneficiary).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged > 60 years with recent fracture (less of 3 months) included in existing FLS in France
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
To compare the efficacy of eFLS to conventional FLS to initiate an antiosteoporotic treatment after a recent fracture (<3 months) at one year in patients aged 60 years and more | one year
  Number of patients receiving an antiosteoporotic treatment at one year

SECONDARY OUTCOMES:
To compare the number of patients with recent fracture (less of 3 months) in the eFLS and conventional FLSs | one year
  Number of patients seen in the FLS
To compare the proportion of patients with incident fracture over one year seen in the eFLS and in conventional FLS | one year
  Incident fracture rate over 1 year
To compare the proportion of patients with deaths over one year in the eFLS and in conventional FLS | one year
  Mortality rate over 1 year
To compare the proportion of patients with bone densitometry performed over one year in the eFLS and in conventional FLS | one year
  Bone densitometry at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Karine BRIOT, MD, PhD, Principal Investigator — APHP
Locations (1):
- Cochin Hospital, Rheumatology Department, Paris, France

IPD SHARING:
Plan to Share IPD: No